CLINICAL TRIAL: NCT01568671
Title: Energy Expenditure Responses to Different Temperatures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 120097; 12-DK-0097
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2025-10-14

CONDITIONS: Obesity; Normal Physiology
Keywords: Adult; Body Composition; Accelerometry; Healthy Volunteers; Thermoregulation; Natural History; Healthy Volunteer; HV
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Healthy older lean white men (Experimental): White men aged 55-75 years with BMI between 18.5 and 25.0 kg/m2
  Interventions: Other: Room temperatures
- Healthy young lean black men (Experimental): Black men aged 18-35 years with BMI between 18.5 and 25.0 kg/m2
  Interventions: Other: Room temperatures
- Healthy young lean white men (Experimental): White men aged 18-35 years with BMI between 18.5 and 25.0 kg/m2
  Interventions: Other: Room temperatures
- Healthy young lean white women (Experimental): White women aged 18-35 years with BMI between 18.5 and 25.0 kg/m2
  Interventions: Other: Room temperatures
- Healthy young white men with obesity (Experimental): White men aged 18-35 years with BMI between 30.0 and 40.0 kg/m2
  Interventions: Other: Room temperatures

INTERVENTIONS:
Other: Room temperatures — Room temperature of metabolic chamber set between 16C and 31C

SUMMARY:
Background:

- The way that the body burns calories is known as energy expenditure. Some studies show that when we are cold, we burn more calories to keep our bodies warm. Brown fat is a special kind of fat that can use energy to keep the body warm. Small animals and infants have been known to have brown fat for many years. Recently, it has been suggested that adult humans also have brown fat. If brown fat becomes active (burns calories) in adult humans when exposed to cold, then these people would tend to burn off more calories and might not gain weight easily. Learning more about the relationship between energy expenditure, brown fat, environmental temperature, and body temperature may help explain why some people become obese and other people do not.

Objectives:

* To better understand how the body burns calories when exposed to different temperatures.
* To study brown fat and how it burns calories in cold temperatures.

Eligibility:

* Healthy men between 18 and 35 or 55 and 75 years of age.
* Healthy women between 18 and 35 years of age.
* To control for ethnicity, participants must be non-Hispanic whites or African Americans.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will stay in the Metabolic Unit of the National Institutes of Health Clinical Center as inpatients for no more than 14 days. The length of the hospital stay will depend on how participants respond to the different study temperatures.
* Every afternoon, participants will walk for 30 minutes on a treadmill. All meals will be provided.
* Participants will stay up to 5 hours per day in a specialized room with different temperature settings. Temperatures will range from about 61 degrees to 88 degrees Fahrenheit. Body temperature, activity, calorie burning, and cold/hot sensations will be monitored. On the study day of the coldest temperature, participants will have an imaging study to look for brown fat activity.
* Participants will be compensated for their time and participation at the end of the study.

DETAILED DESCRIPTION:
Surprisingly little is understood about how the body regulates heat production (energy expenditure, EE) in response to subtle changes in environmental temperature. For example, only recently has it been realized that brown adipose tissue is functional in adult humans. It is plausible that the mechanisms governing heat production contribute to regulation of body weight and thus may be contributing to the current obesity epidemic: even small changes in EE, if not compensated by changes in food intake, can have long-term effects on body weight.

The thermoneutral zone (TNZ) is the environmental temperature range over which EE is at a minimum and does not change with environmental temperature. The lower and upper critical temperatures define the temperature limits of the TNZ. At environmental temperatures below the lower critical temperature, the EE vs. environmental temperature graph is reported to be a straight line with the extrapolated X-axis intercept being the defended body temperature. Some of these parameters are predicted to be different for obese as compared to lean individuals. With the global obesity epidemic coinciding with improved indoor temperature control, a better understanding of the relationship between EE and thermoregulation is desirable.

This protocol has three phases. The first is a pilot in lean males to optimize procedures and establish the feasibility, sensitivity, and behavior of the assays. Second, lean and obese male cohorts will be compared to ensure that the expected differences can be observed. Third, additional variables will be examined, such as age, race, sex, and menstrual phase in women.

Specifically, we will map the resting EE response to environmental temperatures from 16-31 degrees Celsius during inpatient stays in the NIH Metabolic Clinical Research Unit. Each day resting EE will be measured in a room respiration calorimeter with a different environmental temperature (subjects will be blinded as to room temperature). The remainder of each study day will be spent at 23-25 degrees Celsius in the individual patient room.

Standard diet and physical activity will be maintained and body weight will be held stable. Additionally core body and skin temperatures, heart rate and variability, muscle activity by surface electromyography, and thermal comfort and hunger using visual analog scales will be measured.

This study will establish techniques and provide baseline normative data, allowing insight into the mechanisms regulating the EE in humans and how these are affected by obesity. It is envisioned that this study will provide the basis for investigation of the effects of acute and chronic weight change and the effects of drug therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Generally healthy.
* Males between the age greater than or equal to 18 -35 years or between 55-75 years, male orand females between the age 18-35 years.
* Self-reported non-Hispanic and non-Latino Caucasian and African-Americans
* Written informed consent.

EXCLUSION CRITERIA:

* Hypo- or hyper-thyroid (history or TSH >5.0<0.4 miU/L)
* Psychological conditions,such as (but not limited to) claustrophobia, clinical depression, bipolar disorders, that would be incompatible with safe and successful participation in this study
* Weight change >5% in the past 6 months or a trained athlete

Blood pressure greater than 140/90 mmHg or current antihypertensive therapy

* History of cardiovascular disease
* BMI <18.5, between 25.1-29.9, and >40 Kg/m(2)
* Diabetes mellitus (fasting serum glucose > 126 mg/dL)
* Liver disease or ALT serum level greater than two times the laboratory upper limit of normal
* Iron deficiency (Ferritin < 30 mcg/L males, < 15 mcg/L females)
* Abnormal kidney function (eGFR<60 ml/min/1.73m(2))
* History of illicit drug or alcohol abuse within the last 5 years; current use of drugs (by history) or alcohol (CAGE greater than or equal to 2)
* Current use of medications/dietary supplements/alternative therapies known to alter energy metabolism
* Pregnancy/breastfeeding/hormonal contraception or childbirth within the last year
* Perimenopausal (as self-described within two years from onset of amenorrhea or current complaints of hot flashes)
* For pre-menopausal women, irregular periods or polycystic ovarian disease
* Current smoker or user of tobacco products
* Metal implant that prevents subject from being in a MRI scanner.

All subjects will be fully informed of the aims, nature, and risks of the study prior to giving written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-04-24 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Resting energy expenditure | Days 7-13 of inpatient stay
  Resting energy expenditure at the lowest tolerable temperature above basal metabolic rate (%), measured by metabolic chamber

SECONDARY OUTCOMES:
Mean skin temperature | Days 1-14
  Weighted average of skin temperatures measured by iBottons at the chest, upper arm, upper leg, and lower leg

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD underlying the primary results
Supporting Information: Study Protocol, ICF
Time Frame: From the time of publication and available indefinitely
Access Criteria: Data will be shared with qualified investigators who provide a protocol with IRB approval. Data sharing requires a signed data use agreement.

REFERENCES:
- [Background] Nedergaard J, Bengtsson T, Cannon B. Unexpected evidence for active brown adipose tissue in adult humans. Am J Physiol Endocrinol Metab. 2007 Aug;293(2):E444-52. doi: 10.1152/ajpendo.00691.2006. Epub 2007 May 1. PMID 17473055
- [Background] Virtanen KA, Lidell ME, Orava J, Heglind M, Westergren R, Niemi T, Taittonen M, Laine J, Savisto NJ, Enerback S, Nuutila P. Functional brown adipose tissue in healthy adults. N Engl J Med. 2009 Apr 9;360(15):1518-25. doi: 10.1056/NEJMoa0808949. PMID 19357407
- [Background] van Marken Lichtenbelt WD, Vanhommerig JW, Smulders NM, Drossaerts JM, Kemerink GJ, Bouvy ND, Schrauwen P, Teule GJ. Cold-activated brown adipose tissue in healthy men. N Engl J Med. 2009 Apr 9;360(15):1500-8. doi: 10.1056/NEJMoa0808718. PMID 19357405
- [Derived] Ouwerkerk R, Hamimi A, Matta J, Abd-Elmoniem KZ, Eary JF, Abdul Sater Z, Chen KY, Cypess AM, Gharib AM. Proton MR Spectroscopy Measurements of White and Brown Adipose Tissue in Healthy Humans: Relaxation Parameters and Unsaturated Fatty Acids. Radiology. 2021 May;299(2):396-406. doi: 10.1148/radiol.2021202676. Epub 2021 Mar 16. PMID 33724063
- [Derived] Brychta RJ, Huang S, Wang J, Leitner BP, Hattenbach JD, Bell SL, Fletcher LA, Perron Wood R, Idelson CR, Duckworth CJ, McGehee S, Courville AB, Bernstein SB, Reitman ML, Cypess AM, Chen KY. Quantification of the Capacity for Cold-Induced Thermogenesis in Young Men With and Without Obesity. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4865-4878. doi: 10.1210/jc.2019-00728. PMID 31150063
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-DK-0097.html